CLINICAL TRIAL: NCT02838537
Title: TRiptan Use and Serious Vascular Events in Elderly Over 65 Years
Acronym: TRUE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: ANSM-RCAPHM13_0293
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Migraine
Keywords: Triptan; Drug utilization; Elderly; Drug abuse; Cardiovascular disease
MeSH Terms: conditions — Migraine Disorders; Substance-Related Disorders; Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Triptan Arm: Users of triptan defined as at least one recorded dispensing of any drug during the follow up, with no recorded of any of these drugs during the previous 6 months ("new or incident users")
  Interventions: Drug: Exposure to Triptan
- Ergot Arm: Users of ergot derivative defined as at least one recorded dispensing of any drug during the follow up, with no recorded of any of these drugs during the previous 6 months ("new or incident users")
  Interventions: Drug: Exposure to Ergot

INTERVENTIONS:
Drug: Exposure to Triptan
  Groups: Triptan Arm
Drug: Exposure to Ergot
  Groups: Ergot Arm

SUMMARY:
This study will be conducted as a retrospective study of exposed and unexposed cohort of the French population included all beneficiaries aged 65 and older. Exposed patients will be matched to non exposed controls according age, gender and area of residence (ratio 1/4). Two exposed arms and two non exposed control arms will be planned. Triptan arm will be user of triptan defined as at least one recorded dispensing of any drug during the follow up, with no recorded of any of these drugs during the previous 6 months ("new or incident users"). Ergot arm will be user of ergot derivative defined as at least one recorded dispensing of any drug during the follow up, with no recorded of any of these drugs during the previous 6 months ("new or incident users"). This study involved data from the French National Health Insurance Information System (Système National d"Information Inter-Régimes de l"Assurance Maladie ; SNIIRAM) linked with the French hospital discharge database (Programme de Médicalisation des Systèmes d"Informations, PMSI).

* The SNIIRAM is a vast national medico-administrative database representing the most part of the French population, allowing to identify and to describe precisely all medication dispensations (name of drug, date of dispensing and quantity) including triptans and other reimbursed medications.
* The PMSI provides medical information about all patients admitted to hospital in France, including discharge diagnoses encoded according ICD-10, medical procedures and French diagnosis-related groups The research proposed is expected to provide an update and nationally-consolidated estimation of the cardiovascular risk is associated to triptans use in elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and more
* Patients registered in the SNIIR-AM
* To avoid depletion of susceptibles bias, only incident users will be included. Incident users are defined by the lack of reimbursement for triptan (or ergot derivatives) prior six months of the study period.

Exclusion Criteria: no exclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Both exposed cohorts will include all beneficiaries recorded in the SNIIR-AM aged 65 and older, who had an incident dispensation of any triptans (or ergot derivatives) over the study period.
  An incident dispensation is defined by the lack of dispensation for triptan (or ergot derivatives) for the first six months of the study period.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Occurence of the first vascular event leading to a hospitalization within the exposure period following the first dispensation of a triptan. | Up to 4 years

SECONDARY OUTCOMES:
Assessment of the mortality: number of all deaths | Up to 4 years
  Assessment of the deaths, whatever the cause
Assessment of the mortality with an underlying cardiovascular cause occuring in hospital | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assitance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided